CLINICAL TRIAL: NCT05252819
Title: Feasibility of Whole-body MRI for Cancer Surveillance in Children and Young People With Ataxia Telangiectasia
Brief Title: Whole Body MRI for Cancer Surveillance in A-T
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Action for A-T (Unknown); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 21062
Record Dates: First submitted 2022-02-04; First posted 2022-02-23 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Ataxia Telangiectasia
Keywords: Ataxia Telangiectasia; Whole-body MRI; Cancer Surveillance
MeSH Terms: conditions — Ataxia Telangiectasia | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging and an optional blood test — One whole-Body MRI that takes approximately 35minutes One blood test, which it is an optional component at this stage

SUMMARY:
Ataxia Telangiectasia (A-T) is an inherited disorder characterised by cerebellar neurodegeneration, immunodeficiency and respiratory disease. People with A-T have abnormal DNA repair and consequently have an increased risk of cancer. Despite this, current guidelines for management of children and young people with A-T do not include cancer surveillance.

Improvements in MRI technology have allowed whole-body MRI (WB-MRI) scanning with relatively short acquisition times. Currently, WB-MRI protocols are used for diagnosing and monitoring some primary and secondary cancers, including cancer surveillance in people with the Li-Fraumeni syndrome, which is another genetic cancer predisposition syndrome. Therefore, the research team believe that whole-body MRI provides a safe method for cancer surveillance in children and young people with A-T. However, the investigators do not know whether cancer surveillance in children and young people with A-T using whole-body MRI is feasible and desirable.

The research team proposes a feasibility study of MRI-based cancer surveillance with qualitative evaluation of participant experience with the primary aim to establish:

* feasibility of whole-body MRI for cancer surveillance in children and young people with A-T
* views of, and psychological impact on, participants and families / carers participating in whole-body MRI for cancer surveillance.
* feasibility of conducting a formal screening trial in terms of statistical design, sample size, screening interval, comparator arms and international collaboration Completion of this study will provide us with evidence of technical feasibility, very strong evidence of child / family views, a viable formal screening trial design and an engaged international research community, allowing us to proceed to a formal trial establishing the efficacy of a cancer surveillance programme for children and young people with A-T.

DETAILED DESCRIPTION:
Ataxia Telangiectasia (A-T) is an autosomal recessive disorder characterised with cerebellar neurodegeneration, immunodeficiency, respiratory disease and cancer susceptibility (22% by age 20). A-T is a complex disorder caused by mutations in the Ataxia Telangiectasia Mutated (ATM) gene which creates highly unstable ATM protein fragments. In the classical clinical presentation of A-T there is no kinase activity due to the absence of ATM protein. One consequence of this is that cellular DNA-repair pathways are compromised which allows breaks in DNA strands leading to genomic instability and/or cell death. As a result, there is an increase sensitivity to ionizing radiation and elevated cancer risk. Children less than 16 years with classical A-T demonstrate a predisposition to the development of different types of lymphoid cancers (lymphoma and leukaemia). However non-lymphoid tumours can also occur.

The current practice at the United Kingdom Paediatric A-T clinic for cancer surveillance is to perform blood testing, including full blood account, liver function tests and measurement of circulating tumour marker Alpha-fetoprotein. Full blood account can detect an increase white cell count and abnormal white cell populations and therefore, is effective in detecting most types of leukaemia. Elevation of Alpha-Fetoprotein can be a marker of different types of tumours, for example hepatocellular carcinoma and liver metastases, however is also often elevated in people with A-T. Therefore, its use for detecting cancer in A-T is uncertain and not currently evidence-based. The lack of evidence-based guidelines regarding the optimal cancer surveillance strategy in children with A-T could delay the diagnosis and consequently the treatment plan.

Magnetic Resonance Imaging (MRI) technology has progress rapidly since its discovery, making it possible currently to perform whole-body MRI scans with relatively short acquisition times. Presently, whole-body MRI protocols that include diffusion-weighted imaging and structural (T1/Dixon) acquisitions are used for diagnosing and monitoring cancers (sarcomas, metastases and haematological tumours like myeloma). A further advantage of this technique compared to computed tomography is that does not involve radiation, which is important given the elevated radiosensitivity of people with A-T.

The value of whole-body MRI in people with cancer predisposition has been shown in Li-Fraumeni syndrome, syndrome that, like A-T, is associated with increased risk of haematological and solid tumours. Despite the successful results of using a multimodality protocol for cancer surveillance in Li-Fraumeni syndrome, it cannot be assumed that the results will be the same in people with A-T as the also have respiratory and neurological dysfunction that could influence the tolerability and image quality of the MRI scans. Also, the profile of the tumours differs between these two syndromes. To date, the value of whole-body MRI for cancer surveillance in children and young people with A-T has not been demonstrated. It is unknown whether is possible to obtain diagnostic images, and the spectrum of findings (both cancer and non-cancer) that can be detected has not been reported.

In addition to technical considerations, it is vital to understand the perspectives of people affected by A-T regarding cancer surveillance. Participation in a cancer surveillance programme could increase anxiety for both the participant and family, and it is possible that negative psychological aspects could outweigh the perceived benefits or earlier cancer detection. Compared to other screening programmes, it should be noted that these families are already having to deal with a family member with complex progressive chronic disease, and so emotional and psychological capacity to deal with added anxiety may be limited. Hence, it is important to know, before conducting a full scale trial that will inform the current lack of evidence-based guidelines, whether cancer surveillance in children and young people with A-T using whole-body MRI is feasible and desirable.

ELIGIBILITY:
Inclusion Criteria:

* for MRI scan: Confirmed diagnosis of A-T Aged 5 to 18 years Able to undergo MRI scan without sedation or general anaesthetic, after age-appropriate preparation Able to give informed consent (if 16 or older), or have a parent guardian who is able to give informed consent
* for Post-participation interviews or focus group: Participants who underwent the MRI scan Able to give informed consent (if 16 or older), or have a parent guardian who is able to give informed consent Parents / carers of the participants who underwent the MRI scan Participants and / or parents/carers willing to consent
* for Delphi Study: medical professionals who have 3 years post-qualification experience in A-T medical professionals who are currently employed in a clinical area that is related to A-T

Exclusion Criteria:

* Contra-indication to MRI scan

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young people with Ataxia Telangiectesia and their parents / carers from United Kingdom registred in Paediatric A-T clinic in Nottingham.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of whole-body MRI for cancer surveillance in children and young people with A-T | 1 year
  To establish the rate of completion of whole-body MRI protocol
Determine the feasibility of whole-body MRI for cancer surveillance in children and young people with A-T | 1 year
  To establish the duration of scan tolerated (if not full protocol)
Determine the feasibility of whole-body MRI for cancer surveillance in children and young people with A-T | 1 year
  To assess the diagnostic image quality

SECONDARY OUTCOMES:
Identification of concerns/views of the participants and their families/carers | 6 months
  To establish baseline views on whether people with A-T and their families/carers want such a cancer surveillance programme and what the specific concerns are regarding participating in this cancer screening
Documentation of number of abnormal findings on whole-body MRI and blood metrics (when applicable) | 2 year
  To establish the prevalence of cancer and non-cancer abnormalities detected on whole-body MRI in this population
Documentation of the locations of abnormal findings on whole-body MRI | 2 year
  To establish the spectrum of cancer and non-cancer abnormalities detected on whole-body MRI in this population
Description of the type of abnormal findings on whole-body MRI and blood metrics (when applicable) | 2 year
  To establish spectrum of cancer and non-cancer abnormalities detected on whole-body MRI in this population
Rates of recommendations for further investigation based on whole-body MRI and/or blood test findings | 2 years
  To establish the rate of subsequent medical management based on the MRI and blood test (when applicable) findings
Assessment of the psychological impact of the participants and their families/carers throughout the study | 1 year
  To asses the participant/parent (carer) experience in the lead up to, during and after the surveillance MRI and blood test (when applicable), to assess the emotional impact regarding the diagnostic tests waiting times and to establish the emotional and informational support needed during the process of surveillance
Engagement of the international A-T community | 6 months
  To establish the current practice regarding cancer surveillance in children and young people with A-T across international centres.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided